CLINICAL TRIAL: NCT04334863
Title: A Phase I Study of WP1066 in Children With Refractory and Progressive or Recurrent Malignant Brain Tumors (AflacST1901)
Brief Title: WP1066 in Children With Refractory and Progressive or Recurrent Malignant Brain Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: CURE Childhood Cancer, Inc. (Other); Peach Bowl LegACy Fund (Unknown)
Responsible Party: Principal Investigator, Tobey MacDonald, Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00113194
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Brain Tumor; Medulloblastoma; Brain Metastases
Keywords: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms; Medulloblastoma | interventions — WP1066

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- WP1066 (Experimental): There will be 5 groups based on the enrollment timing. The first group of participants will receive the lowest dose level of WP1066. Each subject within a group will receive an assigned dose of the investigational drug. The dose levels are 4, 6, 8 and 16 mg/kg of the investigational drug given twice a day. The first group will receive the lowest dose level, 4mg/kg twice a day, and subsequent groups will escalate to the next higher dose level. All groups will be treated identically, except for the dose of drug administered, with the liquid formulation of the drug.
  Interventions: Drug: WP1066

INTERVENTIONS:
Drug: WP1066 — WP1066 is an analogue of caffeic acid that is a potent inhibitor of p-STAT3.
  It will be taken by mouth 2 times per day on Monday, Wednesday, and Friday of Weeks 1 and 2 of each 28-day cycle.
  Other Names: STAT3 Inhibitor WP1066

SUMMARY:
In this Phase I clinical study, the investigators plan to offer investigational treatment with the novel JAK2/STAT3 inhibitor WP1066 (Moleculin Biotech, Inc.) to pediatric patients with any progressive or recurrent malignant brain tumor that is refractory to standard treatment and is without known cure.

DETAILED DESCRIPTION:
The goal of this clinical research study is to find the highest tolerable dose of WP1066 that can be given to pediatric patients with recurrent (has returned after treatment) cancerous brain tumors or melanoma that has gotten worse and spread to the brain. The safety of this drug will also be studied.

WP1066 is designed to target the STAT3 pathway in cancer cells, which makes these cells divide, increases new blood vessels to the tumor, causes the cancer cells to move throughout the body and brain, and avoids them being detected by the immune system. Targeting this pathway may cause the immune system to kill the cancer cells. The investigators will administer five escalating doses of WP1066, starting at lowest dose currently found to be safe and tolerable in adults.

WP1066 is not FDA approved or commercially available. It is currently being used for research purposes only.

Up to 36 participants will be enrolled in this study. All will take part at Children's Healthcare of Atlanta (CHOA).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed progressive medulloblastoma, malignant glioma or any other recurrent/progressive malignant brain tumor, for which curative measures do not exist. Primary spinal tumors are eligible. DIPG and DMG H3K27M do not require histological confirmation.
* Patients with DIPG and DMG with H3K27M who are post-radiation but have not exhibited tumor progression are also eligible.
* Patients must have previously undergone standard-of-care treatment including surgery, radiation, and/or first line adjuvant chemotherapy prior to the experimental treatment (WP1066).
* Patients must have recovered from the acute treatment related toxicities (defined as < grade 1 if not defined in eligibility criteria) of all prior chemotherapy, immunotherapy or radiotherapy prior to entering this study. There is no upper limit to the number of prior therapies that is allowed.
* Age > 3 to 25 years.
* Karnofsky or Lansky Performance Scale score > 60%.
* Patients must have normal organ and marrow function as defined below:

  * Absolute neutrophil count> 1,000/mcL
  * Platelets> 100,000/mcL
  * Total bilirubin within normal institutional limits
  * AST(SGOT)/ALT(SGPT)< 5 x (<10 x if taking steroids) institutional upper limit of normal
  * creatinine within normal institutional limits for age OR creatinine clearance> 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal.
  * PT/PTT< 1.5 x normal institutional standard
  * Patients with stable seizures (e.g., no seizures for ≥ 14 days and not requiring escalation or addition of anti-epileptic drugs) will be eligible.
  * Signed informed written consent obtained from patient if 18 years of age or older, or from guardian/legal representative if patient is less than 18 years of age

Exclusion Criteria:

* Patients must have received their last dose of known myelosuppressive anticancer therapy at least three (3) weeks prior to study enrollment or at least six (6) weeks if prior nitrosourea.
* Biologic or investigational agent (anti-neoplastic): Patient must have received their last dose of the investigational or biologic agent ≥ 7 days prior to study enrollment. Antibodies: ≥ 21 days must have elapsed from infusion of last dose of antibody, and toxicity related to prior antibody therapy must be recovered to Grade ≤ 1. Agents with prolonged half-lives: At least three half-lives must have elapsed prior to enrollment.
* Immunotherapy: Patient must have completed immunotherapy (e.g. tumor vaccines, oncolytic viruses. etc.) at least 42 days prior to enrollment.
* Radiation: Patients must have had their last fraction of:

  * Craniospinal irradiation ≥ 3 months prior to enrollment.
  * Other substantial bone marrow irradiation ≥ 6 weeks prior to enrollment
  * Local palliative XRT (small port) ≥2 weeks.
* Stem Cell Transplant: Patient must be ≥ 12 weeks since autologous bone marrow/stem cell transplant prior to enrollment.
* Surgery Patients must be fully recovered from all acute effects of prior surgical intervention.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to WP1066.
* The enzymatic metabolism profile of WP1066 is unknown. Patients who are receiving drugs that significantly interact with the CYP450 enzyme(s) are ineligible. However, if they are switched to other medications with a 2-week washout window, they will be eligible. Patients are also excluded if they have been exposed within 7 days of planned first study treatment day to medications that are predominantly CYP2D6, 2C9 or 2C19 substrates, strong inhibitors or inducers, and sensitive substrates of CYP3A4 with narrow therapeutic range.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* No single lesion can be larger than 5 cm in maximal diameter. There may not be clinically significant midline shift or hydrocephalus.
* The effects of WP1066 on the developing human fetus are unknown. Pregnant women are excluded from this study because WP1066 could potentially be teratogenic or have abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with WP1066, breastfeeding should be discontinued if the mother is treated with WP1066. Female subjects of childbearing potential should be willing to use 2 methods of birth control prior to study entry, during the study, and for 2 months after the last dose of the study drug or be surgically sterile. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of WP1066 administration.
* HIV-positive patients receiving combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with WP1066.
* The potential for further hemorrhaging with the use of WP1066 is unknown. It will be at the PIs discretion to enroll a patient who has a small, asymptomatic brain hemorrhage, but patients who have had symptomatic hemorrhages will be excluded.
* Patients requiring escalation of the corticosteroid dose will be excluded, but patients receiving a stable or decreasing dose for at least one week prior to registration will be eligible.
* The cardiac toxicities of WP1066 are unknown. Thus, patients who have a mean QTc interval >450 ms at baseline will be excluded. Concomitant use of agents that prolong the QT interval will be avoided.
* Patients with uncontrolled seizures or seizure requiring escalation or addition of anti-epileptic drugs will be excluded.
* The use of medical cannabis and CBD oil is prohibited during the first 2 cycles of this protocol. Patients must be off cannabis oil for 3 days prior to enrollment

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2020-05-04 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of WP1066 | 28 Days post-intervention
  Maximum tolerated dose (MTD) of WP1066 in pediatric patients with recurrent or refractory and progressive malignant brain tumors for which there is no known treatment with clinical benefit.
  Maximum tolerated dose (MTD) is determined as the dose level at which 0/6 or 1/6 patients experience a dose-limiting toxicity (DLT) with at least 2 patients experiencing DLT at the next higher dose level. DLT is defined as an adverse event or an abnormal laboratory value assessed as being at least possibly related to the investigational agent that occurs during the first 28 days after administration of the first dose of WP1066.
Change in safety and tolerability of WP1066: Maximum tolerated dose (MTD) and Dose limiting toxicities (DLT) | Up to 2 months after the last study drug dose
  The trial will investigate the maximum tolerated dose (MTD) and record the dose limiting toxicities (DLTs) at least possibly related to the investigational drug, as well as all toxicities related or unrelated that occur. MTD is defined as the dose level at which 0/6 or 1/6 subjects experience a DLT with at least 2 subjects experiencing DLT at the next higher dose level. A minimum of 6 subjects must be treated at the MTD. DLT is defined as a graded adverse event or abnormal lab value at least possibly related to the investigational drug that occurred within 28 days after the first dose of the drug was administered. All toxicities will be recorded and graded throughout the study.

SECONDARY OUTCOMES:
Pharmacokinetic of WP1066: Peak plasma concentration (Cmax) | Days 1, 2, 14, and 15 of course 1
  Cmax is the observed maximum plasma concentration following drug administration. Individual plasma concentration-time data for WP1066 will be used to generate pharmacokinetic parameter estimates using both compartmental and non-compartmental methods.
Pharmacokinetic of WP1066: Time to peak concentration (Tmax) | Days 1, 2, 14, and 15 of course 1
  Tmax is the time to reach maximum plasma concentration after single dose administration. Individual plasma concentration-time data for WP1066 will be used to generate pharmacokinetic parameter estimates using both compartmental and non-compartmental methods.
Pharmacokinetic of WP1066: Area Under the Plasma Concentration-time Curve from time zero to 24 hours (AUC0-24) | Days 1, 2, 14, and 15 of course 1
  AUC0-24 is the area under the plasma concentration-time curve from time zero to 24 hours after the start of WP1066 and will be calculated using the linear trapezoidal. Individual plasma concentration-time data for WP1066 will be used to generate pharmacokinetic parameter estimates using both compartmental and non-compartmental methods.
Pharmacokinetic analysis of WP1066: Clearance from plasma (CL) following drug administration | Days 1, 2, 14, and 15 of course 1
  CL is the systemic (or total body) clearance from plasma following WP1066 administration. It will be determined by dose/AUC. Individual plasma concentration-time data for WP1066 will be used to generate pharmacokinetic parameter estimates using both compartmental and non-compartmental methods.
Pharmacokinetic analysis of WP1066: Elimination half life (t1/2) | Days 1, 2, 14, and 15 of course 1
  Elimination half-life (t1/2) will be calculated by 0.693/k. Individual plasma concentration-time data for WP1066 will be used to generate pharmacokinetic parameter estimates using both compartmental and non-compartmental methods.
Pharmacokinetic analysis of WP1066: Apparent volume of distribution | Days 1, 2, 14, and 15 of course 1
  Apparent volume of distribution will be calculated by Cl/k. Individual plasma concentration-time data for WP1066 will be used to generate pharmacokinetic parameter estimates using both compartmental and non-compartmental methods.
Pharmacokinetic analysis of WP1066: change in accumulation ratio of WP1066 | Day 1 of cycle 1 (each cycle is 28 days) and Day 7 of cycle 1
  Accumulation ratio of WP1066 will be calculated as the ratio of AUC0-24 on cycle 1 Day 1 vs Cycle 1 fourth dose. Individual plasma concentration-time data for WP1066 will be used to generate pharmacokinetic parameter estimates using both compartmental and non-compartmental methods.
Pharmacodynamic analysis of WP1066: level of activated Stat3 | Hours 0, 4, 24 of Day 1 and Hours 0, 4, 24 of Day 7
  Activated Stat3 is a transcription factor which in humans is encoded by the STAT3 gene. It is a member of the STAT protein family. The level of activated Stat3 (phospho-Stat3) will be measured in the peripheral blood mononuclear cells (PBMCs), the type of immune cells present in the blood, and the immune cytokines in the serum of subjects pre and post administration of the investigational drug.
Change in overall response rate (ORR) of WP1066 treatment | Up to 2 months after the last study drug dose
  Change in overall response rate (ORR) of WP1066 treatment for this pediatric study population in those with radiographically measurable disease.
Change in Immunological response | Up to 2 months after the last study drug dose
  If clinically indicated and as an optional procedure, biopsy or surgery specimens of the tumors will be obtained to determine the molecular expression of p-STAT3, Ki-67 and immunological characteristics of the tumors (Treg infiltration, co-stimulator molecule expression, etc.)
Time to radiographically assessed progression and/or response to treatment with WP1066. | Up to 2 months post-intervention
  The subjects will undergo imaging at baseline and again within 30 days after obtaining the MRI that aroused the suspicion of progression, or an alternative imaging method can be employed, such as MRI with spectroscopy and/or perfusion, or positron emission tomography (PET).
Change in progression-free survival (PFS) | Up to 2 months after the last study drug dose
  The PFS will be defined radiographically as a greater than 25% increase in tumor volume (in malignant glioma) on T1-weighted MRI scans compared with the MRI obtained within 4 weeks before enrollment.
  Estimated using Kaplan-Meier survival curves. Cox proportional hazards regression methodology may be used to assess the association between duration of response or survival and clinical and demographic characteristics of interest.
Change in overall survival (OS) | Up to 2 months after the last study drug dose
  Estimated using Kaplan-Meier survival curves. Cox proportional hazards regression methodology may be used to assess the association between duration of response or survival and clinical and demographic characteristics of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Tobey MacDonald, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta (CHOA), Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Castellino RC, Mumme HL, Franson AT, Yu B, Robinson MH, Dhodapkar K, Aguilera D, Schniederjan MJ, Keesari R, He Z, Bhasin M, Priebe W, Heimberger AB, MacDonald TJ. First-in-child phase I trial of p-STAT3 inhibitor WP1066 in pediatric brain tumor patients. JCI Insight. 2025 Dec 11:e194823. doi: 10.1172/jci.insight.194823. Online ahead of print. PMID 41379553